CLINICAL TRIAL: NCT01384266
Title: A Randomized, Multicenter, Masked Evaluation of 0.5% Loteprednol Etabonate Versus 1% Prednisolone Acetate for the Treatment of Inflammation Following Cataract Surgery
Brief Title: A Comparison of 0.5% Loteprednol Etabonate Versus 1% Prednisolone Acetate Following Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Associated Eye Care, Minnesota (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Stephen S. Lane, MD, Prinicipal Investigator, Associated Eye Care, Minnesota
Other Study IDs: AEC-001
Record Dates: First submitted 2011-01-13; First posted 2011-06-29 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Intraocular Inflammation
Keywords: Intraocular Inflammation following routine Cataract Surgery
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects undergoing Cataract Surgery: Subjects undergoing routine cataract surgery

SUMMARY:
Patients are routinely given steroid eye drops following cataract surgery. This study will compare 2 approved drops:Loteprednol Etabonate versus Prednisolone Acetate Eye drops used following cataract surgery. Patients will be randomly assigned to one drop or the other, and evaluated for inflammation and intraocular pressure as part of the comparison. The study Doctor will be masked as to which drop the patient receives to avoid bias.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 and older undergoing routine cataract surgery.

Exclusion Criteria:

1. Subjects being treated for elevated intraocular pressure, retinopathy, maculopathy, cornea or vitreous opacities that would interfere with visual acuity.
2. Subjects with diabetes, pseudoexfoliation, uveitis, corneal endothelial disease, or active Herpes Simplex Virus(HSV) or Herpes Zoster Virus(HZV) Pupil Stretch and/or Limbal Relaxing Incision(LRIs) will be allowed.
3. Subjects with previous ocular trauma or intraocular surgery
4. Subjects with sensitivities to steroids.
5. Women who are not post-menopausal or are of child bearing potential will be excluded.
6. Intraoperative complications during surgery including posterior capsule rupture and vitreous loss
7. Subjects with best visual potential in the fellow eye worse than 20/60
8. Subjects who are expected to require concurrent ocular or systemic therapy with non-steroidal anti-inflammatory drugs (NSAIDS) mast cell stabilizers, antihistamines, or decongestants within 2 days prior to or during the 21 days following surgery. (Intraoperative NSAIDS for mydriasis are permitted.) 325 mg Aspirin is permitted.
9. Subjects who are expected to require concurrent ocular or systemic corticosteroids, immunosuppressants (including Restasis) within 14 days prior to or 21 days following surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eye Clinic
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Intraocular inflammation grading | Day 21 Post-op
  Slit Lamp examination will be done at each visit to grade intraocular inflammation

SECONDARY OUTCOMES:
Intraocular pressure spikes | Day 21 post-op
  Intraocular pressure(IOP) will be measured at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Lane, MD, Principal Investigator — Associated Eye Care
Locations (2):
- United States (2):
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Associated Eye Care, Stillwater, Minnesota